CLINICAL TRIAL: NCT03770351
Title: Precision Medicine for Early Prostate Cancer: Integrating Biological and Patient Complexity Variables to Predict Treatment Response
Brief Title: Early Prostate Cancer: Predicting Treatment Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other); Cedars-Sinai Medical Center (Other); VA Medical Center-West Los Angeles (U.S. Federal Agency); VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CIAPM [HS# 2017-3634]
Record Dates: First submitted 2018-12-03; First posted 2018-12-10 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: genomics; racial disparities; patient reported outcomes
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — De-identified specimens stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will replicate/validate the risk prediction model developed for the Comparative Effectiveness Analysis of Surgery and Radiation (CEASAR) study in a more diverse patient population to assess generalizability of the model as well as evaluate the relative contribution of the Decipher Prostate Cancer Test and ProstateNext Test from Ambry Genetics, to the risk prediction model for estimating treatment outcomes, and thereby improve personalization of treatment options.

DETAILED DESCRIPTION:
The study will contribute a replicable model for improving risk prediction from patient characteristics, clinical severity indicators, and genomic tests to aid in personalizing treatment. The proposed registry would also allow future comparisons of the gene expression used in other competing commercial test. The addition of the suggested genomic classifier and its associations with other patient and clinical characteristics will enhance the ability of future studies, analogous to CEASAR, to accurately predict the risk of tumor aggressiveness in prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 90 years of age
* Prostate-Specific Antigen (PSA) values <50ng/ml
* Clinical stage of T1 or T2
* No evidence of metastasis or nodal involvement

Exclusion Criteria:

* Age 91 or greater
* Clinically locally advanced or metastatic disease
* PSA equal to or greater than 50ng/ml
* Diagnosis of malignancy (excluding squamous or basal cell carcinoma of the skin) within 3 years of diagnosis of prostate cancer

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since this study is working with prostate cancer, our cohort will only be males.
Study Population: Our study population will be selected from clinics at 5 major southern California hospitals including: University of California, Irvine, University of California, Los Angeles, Cedars-Sinai Medical Center, Veterans Affair Healthcare Center Long Beach, and Veterans Affair Healthcare Center West Los Angeles.
Sampling Method: Non-Probability Sample
Enrollment: 693 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Prostate-Cancer-specific change in quality of life | Day of enrollment, 6-months, and 12-months after enrollment
  Quality of life is measured by the Expanded Prostate Cancer Index Composite (EPIC). The Expanded Prostate Cancer Index Composite [EPIC] is a validated instrument for measuring disease-specific function/ The domain scores range from 0 to 100, with higher scores representing better function. Patients will be asked to complete the questionnaires during a consultation visit or remotely. EPIC scores will be collected at baseline, 6 month follow up, and at 12 month follow up via the questionnaire. EPIC scores from each time point will then be compared to look at the change in quality of life over the duration of the study.

SECONDARY OUTCOMES:
Recurrence of cancer | EMR data abstraction around the 6-month time point after enrollment
  Recurrence will be recorded from data abstraction from the electronic medical records (EMR).
Complications of treatment | EMR data abstraction around the 6-month time point after enrollment
  Complications of treatment will be measured using general scales for identifying complications and severity (the Clavien system) as well as assessment of a priori identified complications that are known to occur with prostate cancer care. This information will be collected from electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Greenfield, Principal Investigator — University of California, Irvine
Locations (5):
- United States (5):
  - University of California, Irvine, Irvine, California
  - Veterans Affair Long Beach Healthcare System, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Veterans Affair West Los Angeles Healthcare System, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for all primary and secondary outcome measures will be consolidated into one database and be made available to all participating research sites.
Supporting Information: SAP, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access will only be allowed for the principal investigators from each research site.